CLINICAL TRIAL: NCT01454115
Title: Placebo-Controlled, Ascending Single-Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of BMS-708163 in Healthy Male Subjects and a Comparison to Elderly Male and Female Subjects
Brief Title: Study to Evaluate the Safety, Pharmacokinetics and Tolerability of BMS-708163
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CN156-001
Record Dates: First submitted 2011-10-07; First posted 2011-10-18 (Estimated); Last update posted 2011-11-21 (Estimated); Status verified 2011-11

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — BMS 708163

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (14):
- Panel 1: BMS-708163 or Placebo (Experimental): Healthy male subjects (age: 18 to 45 years)
  Interventions: Drug: BMS-708163 (Gamma-Secretase Inhibitor); Drug: Placebo matching BMS-708163
- Panel 2: BMS-708163 or Placebo (Experimental): Healthy male subjects (age: 18 to 45 years)
  Interventions: Drug: BMS-708163 (Gamma-Secretase Inhibitor); Drug: Placebo matching BMS-708163
- Panel 3: BMS-708163 or Placebo (Experimental): Healthy male subjects (age: 18 to 45 years)
  Interventions: Drug: BMS-708163 (Gamma-Secretase Inhibitor); Drug: Placebo matching BMS-708163
- Panel 4: BMS-708163 or Placebo (Experimental): Healthy male subjects (age: 18 to 45 years)
  Interventions: Drug: BMS-708163 (Gamma-Secretase Inhibitor); Drug: Placebo matching BMS-708163
- Panel 5: BMS-708163 or Placebo (Experimental): Healthy male subjects (age: 18 to 45 years).
  In Period 2: Subjects will receive BMS-708163 or placebo as a capsule formulation.
  In Period 3: Subjects will receive BMS-708163 or placebo as a capsule formulation within 5 minutes of consuming a standard high-fat breakfast on Day 1
  Interventions: Drug: BMS-708163 (Gamma-Secretase Inhibitor); Drug: Placebo matching BMS-708163
- Panel 6: BMS-708163 or Placebo (Experimental): Healthy male subjects (age: 18 to 45 years)
  Interventions: Drug: BMS-708163 (Gamma-Secretase Inhibitor); Drug: Placebo matching BMS-708163
- Panel 7: BMS-708163 or Placebo (Experimental): Healthy male subjects (age: 18 to 45 years)
  Interventions: Drug: BMS-708163 (Gamma-Secretase Inhibitor); Drug: Placebo matching BMS-708163
- Panel 8: BMS-708163 or Placebo (Experimental): Healthy male subjects (age: 18 to 45 years)
  Interventions: Drug: BMS-708163 (Gamma-Secretase Inhibitor); Drug: Placebo matching BMS-708163
- Panel 9: BMS-708163 or Placebo (Experimental): Healthy, elderly male subjects (age: 60 years and greater)
  Interventions: Drug: BMS-708163 (Gamma-Secretase Inhibitor); Drug: Placebo matching BMS-708163
- Panel 10: BMS-708163 or Placebo (Experimental): Healthy, elderly female subjects (age: 60 years and greater)
  Interventions: Drug: BMS-708163 (Gamma-Secretase Inhibitor); Drug: Placebo matching BMS-708163
- Panel 11: BMS-708163 or Placebo (Experimental): Healthy male subjects (age: between 46 to 59 years)
  Interventions: Drug: BMS-708163 (Gamma-Secretase Inhibitor); Drug: Placebo matching BMS-708163
- Panel 12: BMS-708163 or Placebo (Experimental): Healthy male and/or female subjects or subjects with MCI (age: between 60-74 years)
  Interventions: Drug: BMS-708163 (Gamma-Secretase Inhibitor); Drug: Placebo matching BMS-708163
- Panel 13: BMS-708163 or Placebo (Experimental): Healthy male and/or female subjects or with AD or MCI (age: 75 years or greater)
  Interventions: Drug: BMS-708163 (Gamma-Secretase Inhibitor); Drug: Placebo matching BMS-708163
- Panel 15: BMS-708163 or Placebo (Experimental): Healthy young male subjects
  Interventions: Drug: BMS-708163 (Gamma-Secretase Inhibitor); Drug: Placebo matching BMS-708163

INTERVENTIONS:
Drug: BMS-708163 (Gamma-Secretase Inhibitor) — Oral Solution, Oral, 0.3 mg, Once daily, once
  Arms: Panel 1: BMS-708163 or Placebo
Drug: BMS-708163 (Gamma-Secretase Inhibitor) — Oral Solution, Oral, 1.5 mg, Once daily, once
  Arms: Panel 2: BMS-708163 or Placebo
Drug: BMS-708163 (Gamma-Secretase Inhibitor) — Oral Solution, Oral, 5.0 mg, Once daily, once
  Arms: Panel 3: BMS-708163 or Placebo
Drug: BMS-708163 (Gamma-Secretase Inhibitor) — Oral Solution, Oral, 15.0 mg, Once daily, once
  Arms: Panel 4: BMS-708163 or Placebo
Drug: BMS-708163 (Gamma-Secretase Inhibitor) — Oral Solution, Oral, 50 mg, Once daily, once
  Arms: Panel 10: BMS-708163 or Placebo; Panel 5: BMS-708163 or Placebo; Panel 9: BMS-708163 or Placebo
Drug: BMS-708163 (Gamma-Secretase Inhibitor) — Oral Solution, Oral, 100 mg, Once daily, once
  Arms: Panel 6: BMS-708163 or Placebo
Drug: BMS-708163 (Gamma-Secretase Inhibitor) — Oral Solution, Oral, 200 mg, Once daily, once
  Arms: Panel 7: BMS-708163 or Placebo
Drug: BMS-708163 (Gamma-Secretase Inhibitor) — Oral Solution, Oral, 400 mg, Once daily, once
  Arms: Panel 8: BMS-708163 or Placebo
Drug: BMS-708163 (Gamma-Secretase Inhibitor) — Capsule, Oral, 50 mg, Once daily, once
  Arms: Panel 11: BMS-708163 or Placebo; Panel 12: BMS-708163 or Placebo; Panel 13: BMS-708163 or Placebo; Panel 5: BMS-708163 or Placebo
Drug: BMS-708163 (Gamma-Secretase Inhibitor) — Oral Solution, Oral, 800 mg, Once daily, once
  Arms: Panel 15: BMS-708163 or Placebo
Drug: Placebo matching BMS-708163 — Oral Solution, Oral, 0 mg, Once daily, once
  Arms: Panel 10: BMS-708163 or Placebo; Panel 15: BMS-708163 or Placebo; Panel 1: BMS-708163 or Placebo; Panel 2: BMS-708163 or Placebo; Panel 3: BMS-708163 or Placebo; Panel 4: BMS-708163 or Placebo; Panel 5: BMS-708163 or Placebo; Panel 6: BMS-708163 or Placebo; Panel 7: BMS-708163 or Placebo; Panel 8: BMS-708163 or Placebo; Panel 9: BMS-708163 or Placebo
Drug: Placebo matching BMS-708163 — Capsule, Oral, 0 mg, Once daily, once
  Arms: Panel 11: BMS-708163 or Placebo; Panel 12: BMS-708163 or Placebo; Panel 13: BMS-708163 or Placebo; Panel 5: BMS-708163 or Placebo

SUMMARY:
The primary objective is to assess the safety and tolerability of a single oral dose of BMS-708163 in healthy young male subjects and in elderly male and female subjects.

ELIGIBILITY:
Inclusion Criteria:

* Panels 1- 8 and Panels 14-15: healthy male subjects between the ages of 18 to 45
* Panels 9 and 10: healthy elderly males and females ages 60 and greater
* Panel 11: healthy males between the ages of 46-59
* Panel 12: males and/or females either healthy or with mild cognitive impairment (MCI) between the ages of 60 and 74
* Panel 13: males and/or females, healthy or with Alzheimer's disease (AD) or MCI that were 75 years of age or greater
* Acceptable medical history, physical examinations, vital signs, electrocardiograms, hemoccult stool tests, and clinical laboratory evaluations

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2007-06; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of Single doses of BMS-708163 in the range of 0.3 to 800 mg in the healthy subjects | Within 28 days of dosing
  Based on adverse event reports and the results of vital sign measurements, ECGs, physical examinations, and clinical laboratory tests

SECONDARY OUTCOMES:
Effects of BMS-708163 on cortisol and QT interval corrected for heart rate | Within 28 days of dosing
Effect of BMS-708163 on thyroid stimulating hormone (TSH), free triiodothyronine (T3), free thyroxine (T4), and lymphocyte subsets | Within 28 days of dosing
Bioavailability of BMS-708163 from a capsule formulation relative to a solution formulation | Within 28 days of dosing
Effect of food on the PK of BMS-708163 administered as a capsule formulation | Within 28 days of dosing
Maximum observed plasma concentration (Cmax) of BMS-708163 | Within 28 days of dosing
Time of maximum observed plasma concentration (Tmax) of BMS-708163 | Within 28 days of dosing
Area under the plasma concentration-time curve from zero to the time of the last quantifiable concentration [AUC(0-T)] of BMS-708163 | Within 28 days of dosing
Area under the plasma concentration-time curve from time zero extrapolated to infinite time [AUC(INF)] of BMS-708163 | Within 28 days of dosing
Plasma half-life (T-HALF) of BMS-708163 | Within 28 days of dosing

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- [Derived] Tong G, Wang JS, Sverdlov O, Huang SP, Slemmon R, Croop R, Castaneda L, Gu H, Wong O, Li H, Berman RM, Smith C, Albright CF, Dockens RC. Multicenter, randomized, double-blind, placebo-controlled, single-ascending dose study of the oral gamma-secretase inhibitor BMS-708163 (Avagacestat): tolerability profile, pharmacokinetic parameters, and pharmacodynamic markers. Clin Ther. 2012 Mar;34(3):654-67. doi: 10.1016/j.clinthera.2012.01.022. Epub 2012 Feb 28. PMID 22381714